CLINICAL TRIAL: NCT03931512
Title: Transcranial Direct Current Stimulation Effects on Motor Learning and Motor Control in Healthy Subjetcs
Brief Title: TDCS Effects on Motor Learning and Motor Control in Healthy Subjetcs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Laura Flix Díez, Physiotherapyst, Msc, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-0022/18
Record Dates: First submitted 2019-04-08; First posted 2019-04-30 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: transcranial direct current stimulation; motor learning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcranial direct current stimulation (Experimental): 20 minutes of transcranial direct current stimulation
  1 mA on bi-hemispheric colocation with cathode on the left M1 and anode on the right M1
  Interventions: Device: transcranial direct current stimularion
- sham transcrial direct current stimulation (Sham Comparator): 20 minutes positioning the electrodes on the scalp. Whith an initial increasing of the current intensity by 10 seconds, until 1mA and a ramp down from 20 seconds to reach zero.
  Interventions: Device: transcranial direct current stimularion

INTERVENTIONS:
Device: transcranial direct current stimularion — aplication of direct current stimulation on the scalp wiht sponge electrodes

SUMMARY:
Clinical Trial with two groups, transcranial direct current stimulation aplication and sham; triple blinded. The protocol is applied 5 consecutive days during the training of a manual dexterity task. Manual dexterity and somatosensory variables are measured pre intervention, post one day of intervention, post 5 days of intervention, and 5 days after finish the intervention.

DETAILED DESCRIPTION:
Clinical Trial with two groups, transcranial direct current stimulation aplication (1 mA ) and sham (ramp up and down of 30 seconds in total) . Bouth interventions will last 20 minutes; at the same time of the aplication bouth are going to train the manual dexterity with Purdue Pegboard Test.

This protocol is applied 5 consecutive days, also it have a follow up of 5 days more.

It is triple blinded. Manual dexterity and somatosensory variables are measured pre intervention, post one day of intervention, post 5 days of intervention, and 5 days after finish the intervention.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* metal or skin lesions on the head
* brain stimulation in the last 6 months
* family history of epilepsy or seizures
* pacemaker or any cardiac involvement
* inability to understand or execute the task
* taking drugs that may influence cognition
* pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in trained manual dexterity of the dominant hand | pre intervention, post one day of intervention, post 5 days of intervention, 5 days after finish the intervention
  One hand manual dexterity is measured with Perdue Pegboard test

SECONDARY OUTCOMES:
Changes in trained manual dexterity of bouth hands | pre intervention, post one day of intervention, post 5 days of intervention, 5 days after finish the intervention
  Two hands dexterity is measured with Perdue Pegboard test
Changes in maximal isometric hand grip force | pre intervention, post one day of intervention, post 5 days of intervention, 5 days after finish the intervention
  Hand grip force is measured with Jamar dinamometer
Sleep Quality | 5 days after finish the intervention
  Pittsburgh Sleep Quality Index
Physical activity | 5 days after finish the intervention
  Long form of the International Physical Activity Questionnaire
Changes in nontrained manual dexterity of the dominant hand | pre intervention, post one day of intervention, post 5 days of intervention, 5 days after finish the intervention
  One hand dexterity is mesured with Minesota Test
Changes in nontrained manual dexterity of bouth hands | pre intervention, post one day of intervention, post 5 days of intervention, 5 days after finish the intervention
  Two hands dexterity is mesured with Minesota Test
Changes in pressure detection treshold | pre intervention, post one day of intervention, post 5 days of intervention, 5 days after finish the intervention
  The pressure detection treshold is measured with an algometer
Changes in pain detection treshold | pre intervention, post one day of intervention, post 5 days of intervention, 5 days after finish the intervention
  The pain detection treshold is measured with an algometer
Changes in two points discrimination | pre intervention, post one day of intervention, post 5 days of intervention, 5 days after finish the intervention
  Two points discrimination is measured with an esthesiometer

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Lerma Lara, PhD, Principal Investigator — University Studies Center La Salle
Locations (1):
- CEULaSalle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The individual praticipant data is going to be anonymized. Also, the participants are going to sing the consent of shareing his personal data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Just before the clinical trial will be ended, and in an unlimited frame of time.
Access Criteria: With resaserches that will need this information for another studies.